CLINICAL TRIAL: NCT04558619
Title: Exploring the Feasibility of a Group Prenatal Program, Kōmmour Prenatal, to Reduce Maternal and Infant Health Disparities Among Marshallese Pacific Islander Women
Brief Title: Exploring the Feasibility of Kōmmour Prenatal to Reduce Maternal and Infant Health Disparities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 261186
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-08

CONDITIONS: Kōmmour Prenatal Among Marshallese Pregnant Women
Keywords: Kōmmour; Prenatal; Marshallese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kōmmour Prenatal (Other)
  Interventions: Behavioral: Kōmmour Prenatal

INTERVENTIONS:
Behavioral: Kōmmour Prenatal — Centering Pregnancy, a group prenatal care model, is a promising intervention that challenges the standard model of one-on-one counseling of prenatal care. The model, is currently implemented at the UAMS, but as of yet to be adapted for Pacific Islanders. Centering Pregnancy replaces the individual prenatal care visit with a group model for obstetrically low-risk women. This model provides substantially more health promotion content than the traditional one-on-one prenatal care model. The intervention occurs from week 14 of pregnancy through birth, following the same same schedule as individual care. Group visits are 90-120 minutes each and follow a unique structured curriculum that incorporates standards of care. In the group setting, credentialed prenatal providers conduct a one-on-one assessment with each patient (30 min) and then facilitate group discussions on the topics of pregnancy, using adult learning principles (60-90 min).

SUMMARY:
The purpose of the study is to culturally adapt and examine the feasibility of a group prenatal program (Kōmmour Prenatal) to reduce maternal and infant health disparities among Marshallese Pacific Islander women in the US. The study will also gather information from providers of Kōmmour Prenatal and stakeholders in the Marshallese community familiar with the program to learn of their experience with the program.

ELIGIBILITY:
Inclusion Criteria

* Women who self-identify as Marshallese
* 18 years of age or older
* And 8-20 weeks pregnant

Exclusion Criteria

* Women who do not self-identify as Marshallese
* Not 18 years of age or older
* And not 8-20 weeks pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Gestational Weight Gain | 9 months
  Gestational weight gain will be measured by weight of first and last group prenatal visit along with information from the birth record data. We will use independent samples tests for proportions to compare treatment groups. We will also use generalized linear models to examine treatment group differences including important covariates such as income, education, age and marital status. Further, data from the proposed study will be use the data from the Kommour treatment group to estimate intraclass correlations as an indicator of clustering due to the nesting of participants within groups.

SECONDARY OUTCOMES:
Breastfeeding initiation, birth weight of infant, preeclampsia, primary cesarean birth, and gestational diabetes mellitus | 9 months
  The research team will abstract medical record information about the mother and child.

CONTACTS AND LOCATIONS:
Overall Officials: Britni Ayers, PhD, Principal Investigator — University of Arkansas for Medical Sciences Northwest
Locations (1):
- University of Arkansas for Medical Sciences Northwest, Fayetteville, Arkansas, United States

REFERENCES:
- [Derived] Ayers BL, Eswaran H, CarlLee S, Reece S, Manning N, McElfish PA. Exploring the feasibility, acceptability, and preliminary effectiveness of a culturally adapted group prenatal program, CenteringPregnancy, to reduce maternal and infant health disparities among Marshallese Pacific Islanders: A study protocol. Contemp Clin Trials Commun. 2023 Apr 3;33:101127. doi: 10.1016/j.conctc.2023.101127. eCollection 2023 Jun. PMID 37091509